CLINICAL TRIAL: NCT04208165
Title: Ultrasound Guided Paravertebral Block Versus Transverse Abdominis Plane Block in Hepatic Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: PVB Versus TAP in Hepatic Patients Undergoing Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Hanan Farouk Khafagy, Professor doctor, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TBRI 118
Record Dates: First submitted 2019-12-14; First posted 2019-12-23 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Ultrasound Therapy; Hepatic Impairment; Laparoscopic Cholecystectomy
Keywords: Ultrasound- guided; PVB; TAP; Hepatic; Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (ultrasound-guided PVB) (Active Comparator): In group P, the patient is in sitting position, a linear transducer (6-15 MHz) placed just lateral to the spinous process. Once the transverse processes and ribs are identified, the transducer is moved slightly cauded into the intercostal space between adjacent ribs to identify the thoracic paravertebral space (PVS) and the adjoining intercostal space. The hyper echoic line of the pleura and underlying hyper echoic air artifacts move with respiration. The needle stimuplex needle will be inserted and 0.5- 1 ml local anesthetic injection administered to show the displacement of pleura downward followed by 15 cc bupivacaine 0.25% into each side the PVS. A pop often is felt as the needle penetrates the internal intercostal membrane. Intravascular injection will be eliminated by negative aspiration before injection. Local anesthetic (15- 20 ml) is slowly injected in small increments, avoiding forceful high-pressure injection to reduce the risk of bilateral epidural spread.
  Interventions: Other: ultrasound-guided nerve block PVB
- Group T (ultrasound-guided TAB) (Active Comparator): In group T, Subcostal blockage will be done in plane technique with 22 G needle (BRAUN Stimuplex D Plus 0,71 50- 80 mm 22 G). The puncture area and the ultrasound probe will be prepared in an aseptic manner. The ultrasound probe is placed in a transverse plane to the lateral abdominal wall in the midaxillary line, between the lower costal margin and iliac crest. On each side, The rectus abdominis and underlying transverses abdominis muscles near the costal margin and xiphoid process will be identified. In-plane image will be obtained and the needle will be inserted through the rectus muscle 2-3 cm medial to the probe. Once the tip of the needle is visualized to be in the plane, 0.25% bupivacaine will be administered incrementally. The drug will be injected along the oblique subcostal line, extending inferolaterally from the xiphoid towards the anterior part of the iliac crest by multiple punctures; a total of 15 ml will be given on each side.
  Interventions: Other: ultrasound-guided nerve block TAB

INTERVENTIONS:
Other: ultrasound-guided nerve block PVB — Thoracic paravertebral block guided by ultrasound device which allows visualizing the surrounding anatomy and placement of the needle at the target location in real time.
  Arms: Group P (ultrasound-guided PVB)
Other: ultrasound-guided nerve block TAB — Transverse abdominis plane block guided by ultrasound device which allows visualizing the surrounding anatomy and placement of the needle at the target location in real time.
  Arms: Group T (ultrasound-guided TAB)

SUMMARY:
The Era of using ultrasound guided blocks provides an attractive and more or less safe alternative to other techniques. Among these blocks is ultrasound-guided transverse abdominis plane block (USG-TAP block) that controls pain by local anesthetic injection into the neurofascial plane of the abdominal muscles. Ultrasound-guided thoracic paravertebral block (USG-TPVB) is another technique in which local anesthetic is injected nearby the thoracic vertebra where spinal nerve emerges from the intervertebral foramina. It provides ipsilateral somatic and sympathetic blockade in many dermatomes around the injection site. The aim of this study is to verify which technique is more efficient in reducing the intra- and postoperative analgesic requirements in hepatic patients.

DETAILED DESCRIPTION:
Study design:

Prospective randomized clinical study, sixty patients will be randomly allocated to one of two groups according to a computer-generated random number table of 30 patients each to receive ultrasound-guided either TAP block (Group T) or PVB (Group P).

Study setting and location Theodor Bilharz research institute.

Study population:

60 patients (ASA II or III ) undergoing laparoscopic cholecystectomy under general anesthesia will be recruited and will be randomly allocated using a computer-generated random number table of 30 patients each to receive either:

1. Paravertebral block group or
2. Transverse abdominis muscle block group.

Study Procedures

Methodology in details :

Anesthesia technique:

Preoperative :

* During the pre-operative period visual analog scale (VAS) for pain assessment from 0 to 10, with 0 meaning no pain and 10 meaning the worst pain imaginable will be explained to patients.
* Midazolam 0.05 mg/kg will be given as pre-medication upon arrival to the operating room then 500 ml lactated Ringer's solution will be administered slowly iv as a pre-load

Monitoring :

ECG, pulse oximetry, noninvasive blood pressure, gas analyzer, bispectral index (BIS), and TOF-Guard module for neuromuscular monitoring (Dragger Infinity Kappa version VF-5W, Germany) are connected to the participants.

Induction and maintenance

* During mask pre-oxygenation, patients' baseline hemo-dynamic parameters will be recorded regarding blood pressure and heart rate.
* General anesthesia will be standardized for all patients with :

1.5- 2 µg / kg fentanyl, 2-2.5 mg/kg 2% propofol then 0.5 mg/kg atracuriam will be administered for muscle relaxation.

* Patients will be intubated and lungs mechanically ventilated to maintain end-tidal CO2 between 30 to 35 mmHg. Fresh gas flow oxygen in air 30-40% at a rate of 3 L/min for 10 minutes will be administered then decreased to 1L/min using a closed system (Fabius GS, Dräger, Lübeck, Germany).
* The patients will receive 1 MAC desflurane which is defined as an expired fraction of 6.0 vol. %. Then the dial-up percentage will be adjusted to establish a BIS value between 40- 50.
* Top- up doses of 0.15 mg/kg atracurium will be given to maintain intra-operative muscle relaxation according to TOF-guard.
* All surgical procedures will be done in the range between 10 am and 2 pm and by the same surgical team.
* Patients will be randomly allocated to one of the 2 groups :

I. In group P, USG-TPVB will be performed with the patient is in sitting position, a linear transducer (6-15 MHz) placed just lateral to the spinous process, the depth of field will be set about 3 cm to start scanning. The transverse processes and ribs will be visualized as hyper echoic structures with acoustic shadowing below them. Once the transverse processes and ribs are identified, the transducer is moved slightly cauded into the intercostal space between adjacent ribs to identify the thoracic para-vertebral space (PVS) and the adjoining intercostal space. The PVS appears as a wedge-shaped hypo echoic layer demarcated by the hyper echoic reflections of the pleura below and the internal intercostal membrane above. It is important to visualize the pleura very clearly at all times. The hyper echoic line of the pleura and underlying hyper echoic air artifacts move with respiration. The needle stimuplex needle (BRAUN Stimuplec D Plus 0,71*50- 80 mm 22 G* 2'', 15°) will be inserted and 0.5 - 1 ml local anesthetic injection administered to show the displacement of pleura downward followed by 15 cc bupivacaine 0.25% Marcaine® flacon, Astra Zeneca, Sweden) into each side the PVS. Visualization of the needle and its tip and controlling its path at all times are essential to avoid inadvertent pleural puncture or entry into the intervertebral foramen. A pop often is felt as the needle penetrates the internal intercostal membrane. Intra-vascular injection will be eliminated by negative aspiration before injection. Local anesthetic (15- 20 ml) is slowly injected in small increments, avoiding forceful high-pressure injection to reduce the risk of bilateral epidural spread.

II. In group T, USG-TAP Subcostal blockage will be done in plane technique with 22 G needle (BRAUN Stimuplex D Plus 0,71 50- 80 mm 22 G). The puncture area and the ultrasound probe will be prepared in an aseptic manner. The ultrasound probe is placed in a transverse plane to the lateral abdominal wall in the midaxillary line, between the lower costal margin and iliac crest. On each side, The rectus abdominis and underlying transverses abdominis muscles near the costal margin and xiphoid process will be identified. In-plane image will be obtained and the needle will be inserted through the rectus muscle 2-3 cm medial to the probe. Once the tip of the needle is visualized to be in the plane, 0.25% bupivacaine will be administered incrementally. The drug will be injected along the oblique subcostal line, extending inferolaterally from the xiphoid towards the anterior part of the iliac crest by multiple punctures; a total of 15 ml will be given on each side.

* When heart rate and blood pressure exceeds 20% of baseline in spite of adequate level of anesthesia guided by BIS, boluses of 0.5 µg/kg fentanyl will be given & the total fentanyl dose will be recorded.
* Atropine 0.5 mg increments will be used to control bradycardia (<50 beat min-1) while hypotension (less than 20% of preanesthetic level) will be managed by increasing fluid infusion rate, decreasing inhalational anesthetic concentration and ephedrine 5 mg.
* Reversal of neuromuscular blockade will be achieved by IV administration of neostigmine 0.05 mg kg-1 and atropine 0.02 mg kg-1.
* Patients will be extubated and transferred to post- anesthetic care unit.

Collected parameters:

Before the operation:

* Age, weight, height, sex, ASA, medical history as well as physical examination will be documented.
* Viral hepatitis markers and liver ultrasonography will be done to verify liver affection.
* The Child-Turcotte-Pugh (CTP) classification including preoperative serum albumin, serum bilirubin, ascites, prothrombin time (PT), or INR (modified CTP score), and grade of encephalopathy will be reported.
* Liver functions AST, ALT and ALP will be taken preoperatively, immediately postoperatively and 24 hours later to rule out any change in liver functions.
* Regarding hemodynamic parameters blood pressure and heart rate will be monitored in each group prior and following the block, induction of general anesthesia as well as endotracheal intubation, then every 10 min till end of the operation.
* The total amount of fentanyl consumption throughout operation will be taken.
* Total anesthetic consumption will also be calculated according to the following formula (18):

Total liquid (ml) = from t=0 to t=end dt The time from the start of end-tidal control (t=0) until the time when the vaporizer will be switched off at the end (t=end).

A conversion factor is detected from the amount of vapor given from each ml of volatile liquid: conversion factor of desflurane is 209 ml calculated from the following formula:

Conversion factor = [density of volatile liquid (g/ml) ×volume at room temperature and pressure (24000 ml)] /molecular weight (g).

Total volatile values used will be calculated by summing the product of usage rate by the duration of each time epoch.

Average volatile usage (ml/h) =

Postoperatively:

* Pain intensity will be estimated by a numeric rating scale (NRS) (0 = no pain, 10 = worst imaginable pain) at rest and on coughing at 2, 4, 6 and 24 hours following the end of surgery. When VAS is exceeding four, boluses of 5 mg intravenous pethidine were given till VAS declined to be less than 4.
* Time to first analgesic demand as well as total analgesic requirements will be recorded.
* Any complications regarding the procedure or the block will be noted as intraperitoneal injection, bowel hematoma and transient nerve palsy as well as Local anesthetic toxicity.
* Length of hospital stay.
* Total amount of analgesia (paracetamol).

ELIGIBILITY:
Inclusion Criteria:

1. Elective laparoscopic cholecystectomy surgery.
2. Age: adult patients between 20 - 65 years old.
3. Gender: Both male and female.
4. ASA Class: II.
5. hepatic patients child A or B

Exclusion Criteria:

1. Refusal of patient.
2. Pregnancy and lactation.
3. Fever or sepsis.
4. Patients ASA class III and IV.
5. Child C hepatic patients
6. Addicts and drug abusers.
7. Patients taking corticosteroids or any cardio - active drugs.
8. Local infection at site of the injection.
9. Allergy to any of the study medications.
10. Severe coagulopathy
11. kyphoscliosis concerning the paravertebral group will be excluded from the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-29 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score | 2 hours after surgery.
  Postoperative pain will be estimated by a numeric rating scale (NRS) (0 = no pain, 10 = worst imaginable pain) on coughing.

SECONDARY OUTCOMES:
Intra-operative fentanyl (analgesic) consumption | During the operation
  The total amount of fentanyl (micro-gram) consumption throughout operation. Fentanyl will be given at induction in a dose 1.5- 2 µg / kg fentanyl. When heart rate and blood pressure exceeds 20% of baseline in spite of adequate anesthesia level, boluses of 0.5 µg/kg fentanyl will be given
Total desflurane (anesthetic) consumption | From start of desflurane application til the end of surgery.
  Amount of consumed desflurane (CC) according to the formula: (Fresh gas flow (liter/min) X vaporizor (%) X1000 )/(Conversion factor) dt.
Postoperative pethidine (analgesic) consumption | 24 hours after operation
  Total amount of pethidine (mg). If NRS is more than 4, boluses of 5 mg intravenous pethidine were given till VAS declined to be less than 4.

CONTACTS AND LOCATIONS:
Overall Officials: Hanan F. Khafagy, Prof., Principal Investigator — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers